CLINICAL TRIAL: NCT02204215
Title: Phase 1 Study of Electric Acupuncture for ICU-acquired Weakness in Mechanical Ventilation Patients With Sepsis/Multiple Organ Dysfunction Syndrome
Brief Title: Electric Acupuncture for ICU-acquired Weakness in Mechanical Ventilation Patients
Acronym: EA-ICUAW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wangxing, Director of Intensive Care Unit, Jiangsu Province Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA-ICUAW
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Failure; Sepsis; Multiple Organ Dysfunction Syndrome
Keywords: Weakness; Mechanical Ventilation; Acupuncture Therapy
MeSH Terms: conditions — Respiratory Insufficiency; Sepsis; Multiple Organ Failure; Asthenia | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electric acupuncture & conservative (Experimental): Electric acupuncture therapy on four limbs 30 min each time, twice per day; or conservative treatment without electric acupuncture.
  Interventions: Device: electric acupuncture; Other: conservative

INTERVENTIONS:
Device: electric acupuncture — Electric acupuncture therapy was made on LI4, LI11, ST36, and ST41 on four limbs for each patient, 30 min for each time, twice per day. Starting from the beginning of mechanical ventilation, to the weaning of the mechanical ventilation.
Other: conservative — General treatment, without electric acupuncture, include passive range-of-motion exercise，q2H turning，minimizing the use of sedation, etc.

SUMMARY:
Intensive care unit acquired weakness (ICU-AW) is common and dramatically affect recovery. The purpose of this study is to determine whether electric acupuncture therapy is effective in the treatment of ICU-AW especially in the patients receiving mechanical ventilation with sepsis or multiorgan system failure.

DETAILED DESCRIPTION:
The principle of acupuncture is to produce bioelectric current, as a consequence, to invigorate the circulation, promote tissue regeneration, relieve pain, enhance the immune function, etc. And electric acupuncture can stimulate bioelectricity activities at acupoints, out of reach for ordinary acupuncture effect, especially in the fields of nerve/muscle recovery and regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sepsis or multiple organ dysfunction syndrome
* Within 48 hours from the initiation of mechanical ventilation

Exclusion Criteria:

* Pregnant patients
* Neuromuscular disease or cerebrovascular accident
* With temporary or permanent pacemaker
* Need to use neuromuscular blocking agents
* Inactivity for more than 5 days before ICU admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
strength related parameters | Participants will be followed until the date of weaning from mechanical ventilation, an expected average of 8 weeks
  muscle force, arm circumference, skin fold thickness

SECONDARY OUTCOMES:
mechanical ventilation duration | Participants will be followed until the date of weaning from mechanical ventilation, an expected average of 8 weeks
  the time span from the beginning of mechanical ventilation, till the weaning of mechanical ventilation
28-day mortality | Participants will be followed until the 28th day after mechanical ventilation
  the mortality till the 28th day after mechanical ventilation
number of participants with adverse events of electric acupuncture | Participants will be followed until the date of weaning from mechanical ventilation, an expected average of 8 weeks
  the adverse enents include fainting, infection, bleeding, viscera damage, and so on.
ICU duration | Participants will be followed until the date of discharge from the ICU, an expected average of 8 weeks
  the time span from the beginning of mechanical ventilation, till the date of discharge from the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Xing Wang, M.D., Principal Investigator — Director of Intensive Care Unit
Locations (1):
- Department of Intensive Care Unit, Jiangsu Province Hospital of TCM, Nanjing, Jiangsu, China